CLINICAL TRIAL: NCT05714566
Title: Research on Biomarkers of Clostridioides Difficile Infection in Inflammatory Bowel Disease Patients Defined by Gut Microbiome and Fecal Metabolomics Alterations
Brief Title: Research on Gut Microbiome and Metabolomics Alterations in C.Difficile Infected IBD Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LY2022-059-B
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Inflammatory Bowel Diseases; Clostridium Difficile Infections; Microtia
Keywords: Inflammatory bowel disease; Clostridium difficile disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Clostridium Infections; Congenital Microtia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IBD
  Interventions: Diagnostic Test: Clostridioides difficile toxin detection
- IBD+CDI
  Interventions: Diagnostic Test: Clostridioides difficile toxin detection
- Health control
  Interventions: Diagnostic Test: Clostridioides difficile toxin detection

INTERVENTIONS:
Diagnostic Test: Clostridioides difficile toxin detection — Using Genexpert kit to detect the stool samples of IBD patients. If C. difficile toxin is positive, the patient is assigned to IBD+CDI group, or else assigned to IBD group. Every sample assigned to Health control group should have negative results for C.difficile toxin tests.

SUMMARY:
The goal of this research is to compare alterations of gut microbiota and fecal metabolomics alterations between inflammatory bowel disease patients infected with or without Clostridioides difficile. The main questions it aim to answer are: which bacterial genus or fecal metabolites can discriminate IBD patients infected or more likely to be infected with Clostridioides difficile and their role in the pathogenesis of Clostridioides difficile.

type of study: observational study participant population/health conditions

1. population diagnosed with Ulcerative colitis or Crohn's disease
2. Having diarrhea Participants will be included in this research. If there is a comparison group: Researchers will compare healthy people without IBD or any diarrhea to see if disease or diarrhea would affect the gut microbiota and metabolites.

ELIGIBILITY:
Inclusion Criteria:

* inpatients diagnosed with ulcerative colitis or Crohn's disease in Renji hospital
* age from 18 to 75 years old

Exclusion Criteria:

* other infection caused diarrhea
* other metabolic diseases or inflammatory diseases
* patients who are not able to send back samples 4-6 weeks after therapy

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. IBD group: inpatients diagnosed with ulcerative colitis or Crohn's disease.
  2. IBD+CDI group: IBD patients positive for C.difficile toxin and having diarrhea
  3. Health control: people without diarrhea or any other intestinal diseases and negative for C.difficile toxin tests
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
C.difficile positive | 1 day
  C.difficile toxin test is positive
C.difficile negative | 1 day
  C.difficile toxin test is negative

CONTACTS AND LOCATIONS:
Overall Officials: Min Li, professor, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai jiaotong university, school of medicine, affliated Renji hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
gut microbiota and metabolites change